CLINICAL TRIAL: NCT04539535
Title: The Effects of a Different Exteroceptive Experience on the Early Motor Repertoire in Infants With Down Syndrome
Brief Title: Infants With Down Syndrome on a Different Surface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Bilge Nur Yardımcı Lokmanoğlu, PT, MSc, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GO 19/581
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Different Surface; Fidgety Movements; General Movements
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Down syndrome (Experimental): We did the General Movements Assessment on standard mattress and experimental mattress in infants with Down syndrome on the same day.
  Interventions: Other: General Movements Assessment on two different surfaces in infants with DS and typically infants on the same day
- Typically infants (Experimental): We did the General Movements Assessment on standard mattress and experimental mattress in typically infants on the same day.
  Interventions: Other: General Movements Assessment on two different surfaces in infants with DS and typically infants on the same day

INTERVENTIONS:
Other: General Movements Assessment on two different surfaces in infants with DS and typically infants on the same day — Different surface

SUMMARY:
This study included infants with Down syndrome who applied to the Faculty of Physical Therapy and Rehabilitation, Developmental and Early Physiotherapy Unit of Hacettepe University. The project is characterized to investigate whether there is any differences on different surface between infants with Down syndrome and typically infants who are in the same conditions.

DETAILED DESCRIPTION:
Down syndrome is the most common chromosomal abnormality among the new-borns and characterized by the cognitive deficits, hypotonia, motor developmental and sensory function problems. The somatosensory system disorder such as touch, proprioception, pain and temperature may be seen in these infants and children. There is a delayed peripheral conduction of the stimulus and delayed cerebral processing may cause the abnormal tactile perception response. In the earliest period of life General Movements (GMs), a gestalt-based observation method is one of the most reliable and valid predictors of neurological dysfunction, and it is widely used. GMs occur in age-specific patterns and are described as fidgety movements between from 3 to 5 months in the post-term age. We did the GMs assessment on two different surfaces in the infants with DS and typically infants on the same day, and therefore assumed that determining the fidgety movements and the concurrent movement would enable to us observe the effect of extroceptive stimulation on the fidgety movements and the concurrent movement.

The aim of this study was to investigate the following questions: (i) are fidgety movements and the concurrent motor repertoire of infants with DS depending on different surfaces?, (ii) do fidgety movements and the concurrent motor repertoire change in neurotypical infants depending on the different surface?, and (iii), what are the differences between infants with DS and neurotypical infants?.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged between 3 and 5 months in both groups
* Infants without any neurological, genetic or metabolic disorder diagnosis in the control group

Exclusion Criteria:

* Infants whose parents did not want to participate study.

Ages: 9 Weeks to 19 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The Prechtl General Movements Assessment | Between 3 - 5 Months
  In the earliest period of life General Movements (GMs), a gestalt-based observation method that is widely used, is one of the most reliable and valid predictors of neurological dysfunction. GMs occur in age-specific patterns and are described as fidgety movements from 3 to 5 months in the post-term age.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Nur Yardımcı Lokmanoğlu, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weijerman ME, van Furth AM, Vonk Noordegraaf A, van Wouwe JP, Broers CJ, Gemke RJ. Prevalence, neonatal characteristics, and first-year mortality of Down syndrome: a national study. J Pediatr. 2008 Jan;152(1):15-9. doi: 10.1016/j.jpeds.2007.09.045. Epub 2007 Nov 19. PMID 18154890
- [Background] Brandt BR. Impaired tactual perception in children with Down's syndrome. Scand J Psychol. 1996 Sep;37(3):312-6. doi: 10.1111/j.1467-9450.1996.tb00663.x. PMID 8857002
- [Background] Einspieler C, Prechtl HF, Ferrari F, Cioni G, Bos AF. The qualitative assessment of general movements in preterm, term and young infants--review of the methodology. Early Hum Dev. 1997 Nov 24;50(1):47-60. doi: 10.1016/s0378-3782(97)00092-3. PMID 9467693
- [Background] Einspieler C, Bos AF, Krieber-Tomantschger M, Alvarado E, Barbosa VM, Bertoncelli N, Burger M, Chorna O, Del Secco S, DeRegnier RA, Huning B, Ko J, Lucaccioni L, Maeda T, Marchi V, Martin E, Morgan C, Mutlu A, Nogolova A, Pansy J, Peyton C, Pokorny FB, Prinsloo LR, Ricci E, Saini L, Scheuchenegger A, Silva CRD, Soloveichick M, Spittle AJ, Toldo M, Utsch F, van Zyl J, Vinals C, Wang J, Yang H, Yardimci-Lokmanoglu BN, Cioni G, Ferrari F, Guzzetta A, Marschik PB. Cerebral Palsy: Early Markers of Clinical Phenotype and Functional Outcome. J Clin Med. 2019 Oct 4;8(10):1616. doi: 10.3390/jcm8101616. PMID 31590221
- [Background] Linkous LW, Stutts RM. Passive tactile stimulation effects on the muscle tone of hypotonic, developmentally delayed young children. Percept Mot Skills. 1990 Dec;71(3 Pt 1):951-4. doi: 10.2466/pms.1990.71.3.951. PMID 1705697